CLINICAL TRIAL: NCT03130543
Title: A Randomized Trial of Thickened Feeds to Treat Gastroesophageal Reflux in Children Admitted to Boston Children's Hospital After Brief Resolved Unexplained Event
Brief Title: A Trial of Thickened Feeds to Treat Gastroesophageal Reflux in Children Admitted After Choking Spell
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Focusing on observational cohort study due to limited enrollment in trial
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Rachel Rosen, Associate Professor of Pediatrics, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00023342
Record Dates: First submitted 2017-03-06; First posted 2017-04-26 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Apparent Life Threatening Event; Gastroesophageal Reflux; Aspiration
Keywords: Brief resolved unexplained event
MeSH Terms: conditions — Brief, Resolved, Unexplained Event; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Formula (No Intervention): This is the group of subjects randomized to receive their standard formula
- Standard Formula with Rice Cereal (Experimental): This is the group of subjects randomized to receive their standard formula with rice cereal added
  Interventions: Dietary Supplement: Rice cereal
- Enfamil AR (Experimental): This is the group of subjects randomized to receive Enfamil AR
  Interventions: Dietary Supplement: Enfamil AR

INTERVENTIONS:
Dietary Supplement: Rice cereal — Standard formula thickened with rice cereal
  Arms: Standard Formula with Rice Cereal
Dietary Supplement: Enfamil AR — Enfamil AR formula
  Arms: Enfamil AR

SUMMARY:
Infants often present to the hospital with episodes of coughing, choking, gagging, change in muscle tone, and/or change in skin color, known as brief resolved unexplained event. Many studies have tried to address why infants have these symptoms and if there is a way to prevent them from happening again. Currently, there is no clear agreement on the most common cause of these symptoms or how to prevent them. Some studies have suggested that gastroesophageal reflux can cause these symptoms. The investigators are conducting a study of infants who are admitted to Boston Children's Hospital with episodes of coughing, choking, gagging, change in muscle tone, and/or change in skin color, symptoms that could be reflux. The investigators want to determine if these symptoms can be prevented by changing the way infants are fed, either by giving them a formula to treat reflux or by thickening their feeds to treat reflux. The goal of the study is to determine if different types of feeding interventions prevent infants from coming back to the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients less than 12 months of age who have been admitted to the hospital after brief resolved unexplained event

Exclusion Criteria:

* Patients with any pre-existing significant medical diagnosis (congenital heart disease, known neurologic impairment with or without seizure disorder, other congenital anomalies)
* Patients with any prior hospitalization for BRUE
* Patients with food allergies such that they cannot be on a milk or rice based diet
* Any patient exclusively breastfed because change to a formula or adding thickening is not possible unless patients choose to pump breast milk and stop all nursing

Ages: 0 Years to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2021-04-02 (Actual)

PRIMARY OUTCOMES:
Choking episodes | 2 weeks
  Frequency of choking episodes

SECONDARY OUTCOMES:
Choking episodes | 12 months
  Frequency of choking episodes
Repeat hospital admission | 12 months
  Number of hospitalizations after randomization
Microbiome changes | 2 months
  Prior studies have suggested that infant thickeners can be associated with necrotizing enterocolitis in infants; the aim of this secondary outcome measure will be to evaluate for changes in microbiome (particularly toward a more pathogenic microbiome) after randomization
Urine concentration | 2 months
  Change in urine concentration after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Rachel L Rosen, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duncan DR, Amirault J, Mitchell PD, Larson K, Rosen RL. Oropharyngeal Dysphagia Is Strongly Correlated With Apparent Life-Threatening Events. J Pediatr Gastroenterol Nutr. 2017 Aug;65(2):168-172. doi: 10.1097/MPG.0000000000001439. PMID 27741062